CLINICAL TRIAL: NCT01667094
Title: Continuous-infusion Anti-pseudomonal β-lactams for the Treatment of Acute, Infective Pulmonary Exacerbations in Cystic Fibrosis
Brief Title: A Study Comparing Continuous Infusion Antibiotics to Standard Treatment for Lung Infections in Cystic Fibrosis
Acronym: CISTIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Katherine Langan, PhD, The Alfred
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 249/12; U1111-1132-8291 (Other: Universal Trial Number)
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis
Keywords: Pulmonary exacerbation; Continuous infusion; Antipseudomonal beta-lactams
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent, short infusion (Active Comparator): Infusion over 30 minutes of either:
  Cefepime 1g q8/24 OR Ceftazidime 2g q8/24 OR Meropenem 1g q8/24 OR Piperacillin-Tazobactam 4.5g q8/24 OR Ticarcillin-clavulanate 3.1g q6/24
  Antibiotic chosen by treating physician
  Interventions: Drug: Intermittent, short infusion Ceftazidime; Drug: Intermittent, short infusion Meropenem; Drug: Intermittent, short infusion Ticarcillin-clavulanate; Drug: Intermittent, short infusion Cefepime; Drug: Intermittent, short infusion Piperacillin tazobactam
- Continuous infusion (Experimental): Continuous infusion of either:
  Cefepime 1.5g over 12h, q12/24 after initial loading dose of 500mg OR Ceftazidime 3g over 12h, q12/24 after initial loading dose 1g OR Meropenem 1.5g over 12h, q12/24 after initial loading dose 500mg OR Piperacillin-tazobactam 13.5g over 24h after initial loading dose 2.25g OR Ticarcillin-clavulanate 12.4g over 24h after initial loading dose 1.55g
  Antibiotic chosen by treating physician
  Interventions: Drug: Continuous infusion Ceftazidime; Drug: Continuous infusion Meropenem; Drug: Continuous infusion Ticarcillin-clavulanate; Drug: Continuous infusion Cefepime; Drug: Continuous infusion Piperacillin tazobactam

INTERVENTIONS:
Drug: Intermittent, short infusion Ceftazidime — Ceftazidime 1g q8/24
  Arms: Intermittent, short infusion
Drug: Continuous infusion Ceftazidime — Ceftazidime loading dose 1g infused over 30mins then 3g infused over 12h q12/24
  Arms: Continuous infusion
Drug: Intermittent, short infusion Meropenem — Meropenem 1g q8/24, infusion over 30 minutes
  Arms: Intermittent, short infusion
Drug: Continuous infusion Meropenem — Meropenem initial loading dose of 500mg infused over 30 minutes followed by 1.5g infused over 12/24, q12/24
  Arms: Continuous infusion
Drug: Intermittent, short infusion Ticarcillin-clavulanate — Ticarcillin/clavulanate 3.1g q6/24
  Arms: Intermittent, short infusion
Drug: Continuous infusion Ticarcillin-clavulanate — Ticarcillin-clavulanate loading dose 1.55g followed by 12.4g infused over 24/24 q24/24
  Arms: Continuous infusion
Drug: Intermittent, short infusion Cefepime — Cefepime 1g q8/24
  Arms: Intermittent, short infusion
Drug: Continuous infusion Cefepime — Cefepime loading dose 500mg followed by 1.5g infused over 12/24, q12/24
  Arms: Continuous infusion
Drug: Continuous infusion Piperacillin tazobactam — Piperacillin tazobactam loading dose of 4.5g infused over 30 minutes followed by 18g infused over 24/24, q24/24
  Arms: Continuous infusion
Drug: Intermittent, short infusion Piperacillin tazobactam — Piperacillin tazobactam 4.5g q6/24
  Arms: Intermittent, short infusion

SUMMARY:
Cystic fibrosis (CF) is an inherited disorder which results in increased thickness of secretions, especially in the lungs. By adulthood, the majority of patients with CF will have a bacteria living in their lungs, called Pseudomonas aeruginosa which can cause lung infections. This usually results in worsening respiratory symptoms and often an acute deterioration in their lung function. They are usually treated with antibiotics that target the Pseudomonas aeruginosa. These antibiotics are typically given as short intravenous infusions several times a day. This study aims to compare the standard method of giving these antibiotics with a different strategy of giving these antibiotics to see if this can improve the outcomes of treatment of these infections and reduce the amount of Pseudomonas aeruginosa in the lungs of these patients. This strategy consists of giving the same antibiotics continuously, to ensure there is always enough antibiotic in the bloodstream and the lung to be able to kill the bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >= 18 years of age,
2. Pseudomonas aeruginosa isolated in sputum within the last 12 months,
3. has an acute infective exacerbation, defined by international standards of 2 or more of the following in the last 2 weeks:

   * change sputum volume or colour,
   * increased cough,
   * increased dyspnoea,
   * increased malaise, fatigue or lethargy,
   * anorexia or weight loss,
   * decrease in pulmonary function by 10% or more, or
   * new radiographic changes

Exclusion Criteria:

1. patients < 18 yrs of age,
2. patients that do not meet the criteria for an acute infective exacerbation,
3. concurrent pulmonary embolism, significant haemoptysis, pneumothorax, or respiratory failure,
4. impaired renal function with an estimated creatinine clearance < 60 mls/min,
5. patients allergic to ß-lactam antibiotics,
6. aminoglycoside contra-indicated,
7. intravenous antibiotics in the last 2 weeks, prior to this admission,
8. received more than 24 hours of intravenous antibiotics in this admission,
9. previous lung transplantation,
10. pregnancy or lactation, or
11. inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Cystic Fibrosis Questionnaire-Revised respiratory component (CFQ-R) respiratory symptom score | Day 0 to Day 14

SECONDARY OUTCOMES:
Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory symptom score | Day 0 to Day 7, Day 0 to Day 28
Lung function testing; Forced volume expired in one second (FEV1) | Day 0 to Day 7, Day 0 to Day 28
C-reactive peptide (CRP) | Day 0 to Day 3
Quantitative bacterial load in sputum (total + Pseudomonas aeruginosa) | Day 0 to Day 3, Day 0 to Day 7
  Measured by PCR.
Time above minimum inhibitory concentration (MIC) | Day 3
Antibiotic stability | Day 3
  For ceftazidime and meropenem, antibiotic levels will be measured from the infusion bag at the beginning and end of the infusion to determine the amount of degradation of these antibiotics.
  The temperature of the infusion bags will be monitored continuously during this time.
Pseudomonas aeruginosa virulence gene determinants | Day 0 to Day 3 and Day 0 to Day 7
  A panel of different previously identified virulence gene determinants for Pseudomonas aeruginosa will be measured by RNA analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Peleg, MBBS, FRACP., Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia